CLINICAL TRIAL: NCT04667559
Title: A Prospective, Multicenter Study to Evaluate the Conformis iTotal Identity Knee Replacement System
Brief Title: A Study to Evaluate the Conformis iTotal Identity Knee Replacement System
Status: Terminated | Type: Observational
Why Stopped: Decision of investigational team
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-001
Record Dates: First submitted 2020-11-09; First posted 2020-12-14 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Conformis iTotal Identity Knee Replacement System — The iTotal® Identity KRS is a tri-compartmental semi-constrained knee prosthesis composed of three components: a Femoral Component, a Tibial Component, and a Patellar Component.Using patient imaging, a patient-specific implant is designed that best meets the geometric and anatomic requirements of the specific patient. The treatment allows for the placement of a cemented metallic device designed from the patient's natural bone geometry. This process allows definition of the shape and size of the femoral and tibial components of the implant, as well as the disposable instrumentation.

SUMMARY:
This is a prospective multicenter study located in the United States. Subjects will be implanted with an iTotal Identity Knee Replacement System and followed for 10 years post implantation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical condition included in the approved Indications For Use for the iTotal Identity CR KRS
* Osteoarthritis, as confirmed by the investigator's assessment of disease status at screening visit that warrants a TKR procedure. Disease status is assessed by Clinical and Radiographic assessment.
* Willingness to participate in the clinical study, to give informed consent, and to attend all follow-up visits
* > 18 years of age with complete development of musculoskeletal structures

Exclusion Criteria:

* Simultaneous bilateral procedure required
* BMI > 40
* Active malignancy (defined as a history of any invasive malignancy - except nonmelanoma skin cancer), unless subject has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years
* Poorly controlled diabetes (defined as HbA1c >7 or Investigator discretion)
* Neuromuscular conditions which prevent subject from participating in study activities
* Active local or systemic infection which precludes TKR procedure
* Immunocompromised in the opinion of the Investigator
* Medically diagnosed fibromyalgia or similar conditions that might impact the subject's ability to differentiate source of pain
* Rheumatoid arthritis or other forms of inflammatory joint disease
* Loss of bone or musculature, osteonecrosis, neuromuscular or vascular compromise in the area of the joint to be operated on, to an extent that the procedure is unjustified
* Diagnosed with or receiving treatment for osteoporosis that is likely to confound results in the opinion of the Investigator
* Other physical disability affecting the hips, spine, or contralateral knee that is likely to confound results in the opinion of the Investigator
* Severe instability due to advanced loss of osteochondral structure
* Prior arthroplasty of the affected knee, including High Tibial Osteotomy (HTO)
* Compromised PCL or collateral ligament
* Severe fixed valgus or varus deformity of >15º
* Extensor lag > 15º
* Fixed flexion contracture ≥ 15º
* Unwilling or unable to comply with study requirements
* Participation in another clinical study which would confound results
* Allergy to any of the implant materials
* Pregnant or planning to become pregnant prior to study TKR procedure (in case of pregnancy after study TKR procedure, eligibility to continue with the protocol will be reviewed)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with clinical condition indicated in the approved Instructions for Use for the Conformis iTotal Identity Knee Replacement System
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Pain and function | 2 years post implantation
  Measured by 2011 Knee Society Clinical Rating Score (objective knee score 0-125, function score 0-100, satisfaction score 0-40, expectation score 0-15 with higher scores meaning better outcome)

SECONDARY OUTCOMES:
Revision rate | Post implantation up to 10 years
Incidence of major procedure-related and device-related complications, including infection rate | Post implantation up to 10 years
Post-operative hip-knee-ankle limb alignment (with 180 degrees being the expected outcome, plus or minus 5 degrees), if long leg x-rays available | Post implantation up to 10 years
Number of patients demonstrating radiographic loosening, radiolucency | Post implantation up to 10 years
  Review of x-rays to subjectively determine evidence of implant disassociation with bone
Length of procedure | Implant procedure from time the patient enters the operating room til time the surgery is complete and patient exits the operating room (up to 6 hours)
Length of hospital stay in hours | Time from patient admission to hospital before surgery til discharge from hospital (up to 72 hours)
blood loss during surgery | Implant procedure from time the patient enters the operating room til time the surgery is complete and patient exits the operating room (up to 6 hours)
blood transfusion rates | Implant procedure from time the patient enters the operating room til time the surgery is complete and patient exits the operating room (up to 6 hours)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Personalized Orthopedic Research Institute, Boynton Beach, Florida
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No